CLINICAL TRIAL: NCT02047487
Title: Docetaxel (T), Cisplatin (P) After Induction Chemotherapy With and Without Cisplatin (P) Concurrent Radiotherapy (X) Plus Bevacizumab (B) Phase II Clinical Study
Brief Title: After Induction Chemotherapy of DP Plus DDP Concurrent Radiotherapy With and Without Bevacizumab Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, zhifei zhao, resident physician, Chinese PLA General Hospital
Other Study IDs: S2013-110-02
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a randomized, open controlled multicenter phase II clinical study. The SPSS statistical software estimation of sample size, selection of the initial treatment of locally advanced head and neck squamous cell carcinoma in 120 patients, such as to achieve the desired results, considering expanding the clinical, according to the proportion of 1:1 were randomly divided into two groups, all patients were taken, docetaxel + cisplatin 2 cycles of induction chemotherapy 、Concurrent chemoradiotherapy（tomotherapy+cisplatin）, The experimental group was added with AVASTIN.

ELIGIBILITY:
Inclusion Criteria:

Men and women are not limited, requirements of ECOG0-2, age 18-70 years old, pathological stage III (NCCN2012), had not received radiotherapy and chemotherapy, expected to survive more than 3 months, the routine testing, were in the normal range, signed the informed consent

Exclusion Criteria:

Do not meet the above criteria; allergic to docetaxel and AVASTIN, or metabolic disorders; associated with gastrointestinal bleeding, perforation and other serious diseases; severe liver disease, kidney disease, respiratory disease or unable to control diabetes, hypertension and other chronic disease; heart disease clinical symptoms; there is peripheral nervous system disorders or have obvious mental disorder and disorders of the central nervous system; active phase >CTCAE2 clinical severe infection; a history of organ transplantation (including bone marrow transplantation of autologous peripheral stem cell transplantation); pregnant, lactating women, women of childbearing age and spouse refused to take effective means of contraception contraception; no legal capacity, continue to influence medical or ethical reasons for who

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pathological diagnosis of head and neck squamous cell carcinoma
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
ORR | three month after ratiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: j x li, doctor, Study Chair — Haidian District Fuxing Road, Beijing No. 28 Department of radiotherapy
Locations (2):
- China (2):
  - PLAGH, Beijing
  - PLA307, Beijing